CLINICAL TRIAL: NCT01319448
Title: Safety and Tolerability of Bi-monthly Intermittent Preventive Treatment With Mefloquine-Artesunate or Sulfadoxine-Pyrimethamine Plus Amodiaquine for Prevention of Malaria and Related Complications in Patients With Sickle Cell Anaemia.
Brief Title: Intermittent Preventive Treatment for Malaria in Patient With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Wellcome Trust (Other); University of Ilorin Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5856
Record Dates: First submitted 2011-03-16; First posted 2011-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Malaria; Sickle Cell Crisis
Keywords: Sickle cell disease; Malaria; Intermittent Preventive Treatment (IPT); prophylaxis
MeSH Terms: conditions — Malaria; Vaso-Occlusive Crises; Anemia, Sickle Cell | interventions — Proguanil; Mefloquine; Artesunate; fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Daily proguanil (Active Comparator): Standard policy of a supply of proguanil tablets to be taken daily
  Interventions: Drug: Proguanil
- IPT with MQ+AS bimonthly (Experimental): Intermittent Preventive Treatment (IPT) consisting of a bimonthly course of treatment with mefloquine-artesunate (MQ+AS)
  Interventions: Drug: mefloquine plus artesunate
- IPT with SP+AQ bimonthly (Experimental): IPT with bimonthly course of treatment with sulfadoxine-pyrimethamine plus amodiaquine (SP+AQ)
  Interventions: Drug: Sulfadoxine-pyrimethamine plus amodiaquine

INTERVENTIONS:
Drug: Proguanil — Proguanil tablets, 1.5mg/kg/day
  Arms: Daily proguanil
Drug: mefloquine plus artesunate — This treatment is given once a day for 3 days. Patients weighing 5-8 kg receive one paediatric tablet per day, those weighing 9-17 kg two paediatric tablets, those weighing 18-29 kg one adult tablet and those weighing 30 kg and two adult tablets.
  Arms: IPT with MQ+AS bimonthly
Drug: Sulfadoxine-pyrimethamine plus amodiaquine — amodiaquine plus sulfadoxine-pyrimethamine supervised at each bimonthly clinic visit (amodiaquine 10mg/kg per day for three days and sulfadoxine-pyrimethamine (25/1.25 mg/kg) on the first day).
  Arms: IPT with SP+AQ bimonthly

SUMMARY:
Malaria prophylaxis is recommended for sickle cell disease patients. In Nigeria, daily proguanil or weekly pyrimethamine are the most commonly prescribed regimens, but the current policy is not effective due to poor compliance and drug resistance. Intermittent treatment with a long acting drug regimen administered under supervision at clinic visits may be more effective. The aim of this trial is to compare the tolerability and acceptability of supervised bimonthly treatment with either sulfadoxine-pyrimethamine plus amodiaquine (SP+AQ) or mefloquine plus artesunate (MQ+AS), with the daily proguanil. Two hundred and seventy patients with sickle cell disease attending the paediatric sickle cell disease clinic in Ilorin hospital who meet the eligibility criteria and have parental consent, will be randomized to one of three prophylactic regimens: daily proguanil, bimonthly sulfadoxine-pyrimethamine plus amodiaquine, or bimonthly mefloquine plus artesunate. Patients will be asked to return to clinic every two months and whenever they are sick. At enrollment, the study paediatrician will conduct a physical examination of the child, and collect a venous blood sample for a complete blood cell count and biochemical screen, determination of G6PD genotype, preparation of blood smears for malaria microscopy and a blood spot for determination of molecular markers of resistance. Four days after each clinic visit, patients will be interviewed (by phone and, for a subset, at home or in the clinic) to ask about compliance and adverse events. Participants will be followed for one year. The parents or carer will be encouraged to bring their child to the Outpatient Department clinic if the child becomes unwell. The primary outcome of the trial is tolerability, secondary outcomes are adherence to the regimen, and incidence of malaria and the number of hospitalizations over 12 months. If the bimonthly regimens are well tolerated and the preliminary data from this study are promising, a larger multicentre trial will be required to determine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 6months or older and >=5kg
* Sickle cell clinic attendant
* Both males and females
* Agree to abide by the study protocol
* Give informed consent and assent
* Not acutely sick at the time of recruitment
* Not having additional chronic disease
* Hb genotype of SS and SC confirmed by electrophoresis

Exclusion Criteria:

* known allergy to any of the antimalarial drugs use in the trial,
* severe illnesses requiring urgent admission,
* treatment with sulfadoxine-pyrimethamine or mefloquine in the previous 2wks
* patients on cotrimoxazole prophylaxis

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months
Adherence to the recommended regimen | 12 months

SECONDARY OUTCOMES:
Efficacy against malaria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Milligan, PhD, Study Chair — London School of Hygiene and Tropical Medicine; Kalifa Bojang, PhD, Study Director — MRC Laboratories; Rasaq Olaosebikan, MD, Principal Investigator — University of Ilorin
Locations (1):
- Department of Paediatrics and Child Health, University of Ilorin Teaching Hospital, Ilorin, Kwara State, Nigeria

REFERENCES:
- [Derived] Olaosebikan R, Ernest K, Bojang K, Mokuolu O, Rehman AM, Affara M, Nwakanma D, Kiechel JR, Ogunkunle T, Olagunju T, Murtala R, Omefe P, Lambe T, Bello S, Ibrahim O, Olorunsola B, Ojuawo A, Greenwood B, Milligan P. A Randomized Trial to Compare the Safety, Tolerability, and Effectiveness of 3 Antimalarial Regimens for the Prevention of Malaria in Nigerian Patients With Sickle Cell Disease. J Infect Dis. 2015 Aug 15;212(4):617-25. doi: 10.1093/infdis/jiv093. Epub 2015 Feb 20. PMID 25701866